CLINICAL TRIAL: NCT02448277
Title: A Comparson Among the Use of Direct Laryngoscope.AirwayScope and GlideScope in General Anesthetized Patients Who Require Nasal Endotracheal Tube Intubation
Brief Title: Comparison of Different Tools Inserted Nasal Endotracheal Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB-990188
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2011-04

CONDITIONS: Intubation, Nasotracheal Intubation
Keywords: Macintosh laryngoscope, Pentax, Glidescope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Macintosh Laryngoscope (Experimental): experimental Macintosh Laryngoscope group: laryngoscope is used to assist for nasotracheal intubation.
  Interventions: Device: Macintosh Laryngoscope
- Pentax Airway scope (Experimental): experimental Pentax Airway scope group:Pentax Airway scope is used to assist for nasotracheal intubation.
  Interventions: Device: Pentax Airway scope
- Glidescope (Experimental): experimental Glidescope group:Glidescope is used to assist nasotracheal tube into trachea
  Interventions: Device: Glidescope

INTERVENTIONS:
Device: Macintosh Laryngoscope — the device is to assist nasotracheal intubation
  Other Names: Macintoish laryngoscope
  Arms: Macintosh Laryngoscope
Device: Pentax Airway scope — the device is to assist the nasotracheal tube into trachea
  Arms: Pentax Airway scope
Device: Glidescope — the device is to assist the nasotracheal tube into trachea
  Arms: Glidescope

SUMMARY:
Nasotracheal intubation (NTI) is usually required in patients undergoing maxillofacial surgery. Though video-scopes have been demonstrated to well perform in oral endotracheal intubation, limited information presents in NTI. The aim of the study is to compare the efficacy of video-scopes in NTI and compared with the traditional direct laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists physical status I-III
* aged 20-65 years
* Requiring Nasotracheal Intubation under general anesthesia

Exclusion Criteria:

* mouth open < 3 cm
* limited neck extension < 25 degree
* Ankylosing arthritis patients.
* BMI≧35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
number of the patients with successful nasotracheal intubation and scoring difficult intubation scale | half an hour
  Nasotracheal intubation assisted by a video-stylet may be performed in patients following induction of anesthesia (fentanyl 2 micro-gram/kg, thiamylal 5 mg/kg, cis-atracurium 0.2 mg/kg and propofol 1 mg/kg)

SECONDARY OUTCOMES:
time to intubate | 10 minutes
  time of Intubating the nasotracheal tube (NT) from selected nostril to trachea is continuously calculated but separately into two parts. part one: from termination of mask ventilation and mask removed from face, to the NT tip on the nasopharynx. part two: advancing NT from nasopharynx, through vocal cord into trachea, to present of 3 end tidal carbon dioxide waveforms.

OTHER OUTCOMES:
postoperative nasal bleeding, sore throat and hoarseness | 2 days
  Events of intubating related nasal bleeding are recorded on selected nostril and oral cavity at 3 minutes post-intubation and post-operatively. Incidences of sore throat and hoarseness are evaluated before patients out of recovery room and the following morning

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Yi Tseng, M.D., Study Director — Department of anesthesiology, Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan